CLINICAL TRIAL: NCT04138862
Title: The Reduced Calorie Food and Mood Study: Using Sensory Cues to Optimise the Satiety Value of a Reduced-calorie 'Healthier Choice' Product
Brief Title: The Reduced Calorie Food and Mood Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Keri McCrickerd, Senior Research Fellow, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017/01013
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Markedly Reduced Food Intake; Satiety and Food Intake
MeSH Terms: interventions — Product Labeling

STUDY DESIGN:
Intervention Model Description: Mixed Design:
  4 x Beverage Contexts (assessed in parallel to reduce demand awareness) 2 x Energy Density (assessed as full crossover)
Who Masked: Participant
Masking Description: Single Blind (participant unaware of the meal manipulations)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sensory Matched/Unlabelled (Active Comparator): Sensory-matched covert calorie reduction, unlabelled
  Interventions: Behavioral: Product Labelling and Sensory modifications
- Sensory Matched/Labelled (Experimental): Sensory-matched explicit calorie reduction, labelled
  Interventions: Behavioral: Product Labelling and Sensory modifications
- Sensory Reduced/Labelled (Experimental): Sensory-reduced explicit calorie reduction, labelled
  Interventions: Behavioral: Product Labelling and Sensory modifications
- Sensory Enhanced/Labelled (Experimental): Sensory-enhanced explicit calorie reduction, labelled
  Interventions: Behavioral: Product Labelling and Sensory modifications

INTERVENTIONS:
Behavioral: Product Labelling and Sensory modifications — the beverages varied in the label that was attached (no label or a 'Healthier Choice' label) and the sensory matching of the calorie reduction (sensory matched, reduced or enhanced).

SUMMARY:
Health- and nutrient-related labelling is often used to draw consumer's attention to the potential benefits of consuming one product over another. However, research suggests that products believed to be 'healthier' and/or lower calorie are often experienced as less satiating, and may actually prompt people to consume more or these foods, or others.

The current research aimed to whether consuming a reduced-calorie product labelled "Healthier Choice" affects compensatory eating behaviour (relative to an unlabelled product), and the extent to which this depends on the product's sensory characteristics.

A two-session randomised study was used to test the satiety value of a reduced-calorie beverage - characterised as changes in rated appetite and later food intake (kcal) relative to an original-calorie version - consumed in one of four contexts varying in label and sensory cues. The beverage-contexts were assessed in a non-crossover manner.

DETAILED DESCRIPTION:
Reformulation strategies to reduce the energy density of commonly consumed food and beverage products are needed to support weight management, but one concern is that awareness of consuming 'healthier' foods can promote compensatory eating behaviours. An alternative solution is not to label calorie-reductions so consumers are unaware that they are consuming fewer calories in reformulated products, which has been described as a 'stealth health' approach.

This study investigated whether consuming a reduced-calorie product labelled with Singapore's 'Healthier Choice Symbol' impacts its satiating power relative to an unlabelled control, and the extent to which this can be further modified by changes to the product's sensory characteristics.

Participants were randomised to consume an original (211 kcal per portion; kcal/g) and reduced calorie (98 kcal per portion; kcal/g) versions of a soymilk, with the reduced calorie version presented in one of four beverage context conditions:

* Context 1 - Sensory-matched, unlabelled calorie reduction (control) - Sensory matched to taste like the original (equally sweet, thick and creamy), without a label identifier (covert energy reduction).
* Context 2 - Sensory-matched, labelled calorie reduction - The same sensory matched beverage as above, but with the HCS attached (explicit energy reduction).
* Context 3 - Sensory-reduced, labelled calorie reduction - Designed to taste less thick, sweet and creamy than the original, with the HCS attached (explicit energy reduction).
* Context 4 - Sensory-enhanced, labelled calorie reduction - Designed to taste thicker, creamier and sweeter than the original, with the HCS attached (explicit energy reduction).

Participants consumed the two beverages (original vs. reduced energy) in one of the four beverage contexts on two non-consecutive test sessions at the Clinical Nutrition Research Centre, with at least three days washout between each session. The calorie reduction was conducted as full-crossover while the beverage context groups were assigned non-crossover, to reduce demand awareness.

The primary objective was to assess changes in lunch energy intake (kcal) after consuming the original and reduced-calorie beverages, depending on the beverage context the reduced calorie version was presented in.

The secondary objectives were to assess the sensory evaluations of the beverages (liking and perceived thickness, sweetness and expected fullness etc.), changes in rated appetite up to 180 minutes post-consumption and energy intake (kcal) for the rest of the test day (recorded in a food diary), as a function of the beverages energy density and context.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 and 50 years
* English Speaking

Exclusion Criteria:

* People who are taking insulin or medications known to affect glucose metabolism, appetite or energy metabolism
* Individuals who are currently following a diet program
* People with intolerances or allergies to study foods or test products, e.g. soya, wheat, gluten, cereal, fruits, biscuits, dairy products, rice, vegetable, meat, seafood, sugar and sweetener, gelatin, natural food colourings or flavourings, etc
* Pregnant women
* Regular smokers (> 5 cigarettes per week)
* Individuals with body mass index (BMI) < 18.5 and > 30.0 kg/m2

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Ad libitum intake of a later lunch meal (calories - kcal) | Measured once for up to 20 minutes
  The weight of the test meal consumed during the test session was measured. - There are four test sessions and participants eat one of the four test meals each session. The amount consumed was measured each time.

SECONDARY OUTCOMES:
Changes in rated appetite pre- to post beverage and up to 180 minutes post-consumption, all prior to consuming an ad libitum lunch | pre-meal, immediately post-meal, +15 minutes, +30 minutes, +45 minutes, +60 minutes, +75 minutes, + 90 minutes, + 120 mins, + 150 mins + 180 mins
  100-point Visual Analogue Scale (VAS) ratings of hunger, fullness, desire to eat, prospective consumption and thirst.
Sensory ratings after the first sip of the test beverage | Measured once upon first tasting the test beverage for up to 5 minute
  100-point Visual Analogue Scale (VAS) ratings of thick, sweet, liking, creamy, chalky and sour.
Energy intake (kcal) for across the test day recorded in a Food diary | Up to 24 hours
  Food intake recorded in a food diary and analysed by a trained research assistant using FoodWorks 8.0.3553.

CONTACTS AND LOCATIONS:
Overall Officials: Keri McCrickerd, PhD, Principal Investigator — Clinical Nutrition Research Centre
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No